CLINICAL TRIAL: NCT06994845
Title: A Single-arm, Multicenter, Phase III Study to Assess Efficacy, Pharmacokinetics, Safety and Tolerability of Iptacopan in Pediatric Patients of 2 to <18 Years of Age With Primary Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study to Assess the Efficacy, Pharmacokinetics, Safety and Tolerability of Iptacopan in Pediatric Patients With Primary IgAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLNP023G12301
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Immunoglobulin A Nephropathy (IgAN)
Keywords: Iptacopan,; primary IgA nephropathy,; IgAN,; proteinuria,; UPCR,; eGFR,; kidney function decline,; pediatric,; adolescents
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria | interventions — iptacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- iptacopan (Experimental): Participants in Cohort 1 (12 to < 18 years old) will receive iptacopan at the dose of 200 mg twice per day. Participants in Cohort 2 (2 to < 12 years old) will receive iptacopan at a dose tbd.
  Interventions: Drug: iptacopan

INTERVENTIONS:
Drug: iptacopan — Cohort 1 (12 to < 18 years of age): Iptacopan 200 mg b.i.d.(twice daily) Cohort 2 (2 to < 12 years old): Dosing tbd
  Other Names: LNP023

SUMMARY:
The study is an open-label, single arm, multicenter, Phase III study to determine proteinuria reduction, pharmacokinetics (PK), safety and tolerability (including CV surveillance) of iptacopan in primary immunoglobulin A nephropathy (IgAN) pediatric patients aged 2 to <18 years.

DETAILED DESCRIPTION:
The study will enroll approximately 34 pediatric patients with a diagnosis of primary IgAN by kidney biopsy performed within 3 years of Screening with < 50% tubulointerstitial fibrosis and <25% crescents and not previously treated with immunosuppressive or other immunomodulatory agents within 90 days (or 180 days for rituximab) prior to first study drug administration.

The study comprises the following periods:

* Screening Period (up to 11 weeks)
* Run-in Period (2 weeks): This period will be approximately 14 days prior to the Enrollment Visit (Day 1) to obtain Baseline assessments, including two UPCR FMV measurements (required prior to Day 1).
* Treatment Period ( 52 weeks): The study will enroll approximately 34 pediatric patients in a staggered manner. The approach will be to first enroll Cohort 1 (12 to < 18 years of age) to collect safety data (including CV surveillance data), tolerability data, PK data and biomarker data for up to 52 weeks (EOS). Cohort 1 participants will be enrolled in a single group of 22 participants. Cohort 2 (2 to < 12 years of age) participants will be enrolled in 2 groups with a total 12 participants.
* Follow-up Period (1 week): Participants who completed the Week 52 (EOS) visit and meet all the eligibility criteria may be enrolled in a rollover extension program (REP) in which they will receive open-label iptacopan. Participants who do not enroll in the REP or do not complete Day 1 of the REP within 7 days of the EOS, should be contacted 7 days after the EOS visit for AE and SAE monitoring and any AEs reported by the participant should be recorded in the study case report form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 2 to < 18 years of age as of Day 1.
* eGFR ≥ 30 mL/min/1.73m2 where eGFR is calculated using the modified Schwartz formula at Screening and confirmed during the Run-in Period.
* Kidney biopsy-proven primary IgAN*, with biopsy performed within 3 years of Screening with < 50% tubulointerstitial fibrosis and < 25% crescents. In case a kidney biopsy within 3 years from Screening is not available, a kidney biopsy may be performed if it is part of the planned diagnostic approach and clinical management of the participant.

  * Note: Primary IgAN is defined as any IgAN that is proven by biopsy showing IgA deposits prevalent over the other classes of immunoglobulins and deemed not to be associated with causes of secondary IgAN as per clinical judgment of the Investigator.
* The minimum body weight for participants in Cohort 1 is 35 kg at Screening and confirmed at Baseline (Day 1).
* Proteinuria due to primary diagnosis of IgAN as assessed by UPCR ≥ 1 g/g (113 mg/mmoL) sampled from FMV at Screening on Day -90 and Day -60 as well as during the Run-in Period despite treatment with maximum tolerated dose of ACE inhibitor/ARB for at least 120 days prior to Day 1. Note: UPCR will be assessed based on one FMV sample at Day -90 and based on the geometric mean of 2 FMV samples for the Day -60 visit and during the Run-in Period.
* Vaccination against Neisseria meningitidis and Streptococcus pneumoniae infection is required prior to the start of study treatment. If the participant has not been previously vaccinated, or if a booster is required, vaccine should be given according to local guidelines at least 2 weeks prior to first study drug administration. If study treatment has to start earlier than 2 weeks post vaccination, prophylactic antibiotic treatment should be initiated.
* Vaccination against Haemophilus influenzae is recommended, according to local guidelines, at least 2 weeks before iptacopan.
* All participants must have been on supportive care including stable dose regimen of ACE inhibitor or ARB at either the locally approved maximal daily dose per body weight, or the maximally tolerated dose (per Investigator's judgment for pediatric use), for at least 120 days before first study drug administration. In addition, if participants are taking diuretics, other antihypertensive medication, or other background medication for IgAN (such as SGLT2 inhibitors), the doses should also be stabilized for at least 120 days prior to the first dosing of study treatment.

Exclusion Criteria:

* Any secondary IgAN observed at Screening (and confirmed at Baseline/Day 1) as defined by the Investigator; secondary IgAN can be associated with cirrhosis, celiac disease, human immunodeficiency virus (HIV) infection, herpes simplex virus infection, dermatitis herpetiformis, seronegative arthritis, small-cell carcinoma, lymphoma, disseminated tuberculosis, bronchiolitis obliterans, inflammatory bowel disease, and familial mediterranean fever.
* A clinical diagnosis of immunoglobulin A vasculitis (IgAV or Henoch-Schonlein purpura) based on typical palpable purpura with or without arthralgia and abdominal pain.
* Evidence of significant urinary obstruction or difficulty in voiding at Screening (and confirmed at Baseline/Day 1); any urinary tract disorder or any chronic kidney disease other than IgAN at Screening and before first study drug administration.
* Current acute kidney injury (AKI) defined by Acute Kidney Injury Network (AKIN) criteria within 4 weeks of screening.
* Presence of rapidly progressive glomerulonephritis (RPGN) as defined by 50% decline in eGFR within 3 months prior to Screening or during the Screening and Run-in periods.
* Presence of nephrotic syndrome at Screening based on the investigator's judgment.
* History or current diagnosis of ECG abnormalities indicating significant risk for study participants such clinically significant cardiac arrhythmias, e.g. sustained ventricular tachycardia, or clinically significant second- or third-degree atrioventricular (AV) block without a pacemaker.
* History or current diagnosis of clinically significant echocardiogram abnormalities indicating significant risk for study participants including but not limited to clinically significant functional, morphological and/or structural abnormalities, which may include left ventricular ejection fraction < 50% and/or left ventricular hypertrophy due to uncontrolled blood pressure at Screening.
* Participants of 12 to < 18 years of age with systolic blood pressure (SBP) < 80 mmHg or > 150 mmHg, or diastolic blood pressure (DBP) < 50 mmHg or > 95 mmHg, or pulse rate < 50 bpm or > 110 bpm; participants of 6 to < 12 years of age with SBP < 70 mmHg or > 140 mmHg, or DBP < 40 mmHg or > 90 mmHg or pulse rate < 52 bpm or > 156 bpm; participants of 2 to < 6 years of age with SBP < 70 mmHg or > 120 mmHg, or DBP < 40 mmHg or > 80 mmHg or pulse rate < 52 bpm or > 156 bpm at Screening.
* Participants previously treated with immunosuppressive or other immunomodulatory agents such as but not limited to cyclophosphamide, rituximab, infliximab, canakinumab, mycophenolate mofetil (MMF) or mycophenolate sodium (MPS), calcineurin inhibitors, complement inhibitors (other than iptacopan), oral budesonide, systemic corticosteroids exposure (≥ 0.5 mg/kg/day of prednisone/prednisolone equivalent or > 7.5 mg/d prednisone/prednisolone equivalent total exposure in a single day) within 120 days (or 180 days for rituximab) prior to first study drug administration. Participants treated with endothelin (receptor) antagonists (including sparsentan) within 120 days prior to first study drug administration.
* All transplanted participants (any solid organ transplantation, including bone marrow transplantation).
* History of recurrent invasive infections caused by encapsulated organisms, such as meningococcus and pneumococcus.
* Major concurrent comorbidities at Screening including but not limited to advanced cardiac disease (e.g. New York Heart Association (NYHA) class III (for 6 to <18 years of age), Ross class III (for 2 to < 6 years of age), severe pulmonary disease (e.g. World Health Organization (WHO) class III (for 17 years of age); Pulmonary Vascular Research Institute (PVRI) class III (for 2 to < 17 years of age), or hepatic disease (e.g. active hepatitis) that in the opinion of the investigator precludes participation in the study.
* Current use of any homeopathic and/or herbal medications for IgAN disease progression, such as but not limited to Lei Gong Teng at Screening (and confirmed at Baseline/Day 1).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2030-06-28 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Log-transformed ratio to Baseline in UPCR (based on FMV) | Baseline, Week 38
  UPCR is measured based on the geometric mean of 2 FMVs obtained preceding each scheduled visit.

SECONDARY OUTCOMES:
Pharmacokinetic Parameter Cmax in Plasma | Week 12 (Pre-dose (0), 2, 4, 6, and 8 hours post-dose)
  Cmax is the maximum (peak) observed plasma drug concentration after dose administration (mass x volume-1)
Pharmacokinetic Parameter AUClast in Plasma | Week 12 (Pre-dose (0), 2, 4, 6, and 8 hours post-dose)
  AUClast is the AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1)
Pharmacokinetic Parameter AUCtau in Plasma | Week 12 (Pre-dose (0), 2, 4, 6, and 8 hours post-dose)
  AUCtau is the AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1)
Ctrough concentrations | Week 4, Week 12 and Week 38
  Pre-dose drug concentration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (3):
  - Childrens Hospital Colorado, Aurora, Colorado
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Prim Childrens Hosp Inv Pharm, Salt Lake City, Utah
- Novartis Investigative Site, Nedlands, Western Australia, Australia
- Novartis Investigative Site, Beijing, China
- Israel (4):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
- Novartis Investigative Site, Fuchū, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com